CLINICAL TRIAL: NCT04639141
Title: The Utility of a Synbiotic With Adjunct Gut-directed Hypnotherapy on the Severity of Gastrointestinal Symptoms in Children With Autism
Brief Title: Combined Gut-brain Therapy for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASD-MGB-RCT2020
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder; Functional Gastrointestinal Disorders; Neurodevelopmental Disorders; Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Gastrointestinal Diseases; Neurodevelopmental Disorders; Anxiety Disorders | interventions — Synbiotics

STUDY DESIGN:
Intervention Model Description: Participants will be recruited and randomised (1:1) to one of two 12-week treatment intervention groups: 1) synbiotic or 2) synbiotic + gut-directed hypnotherapy. Follow-up will occur at week 24.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic (Active Comparator): Dosing: one sachet/dose per day for 12 weeks. The combination includes: Lactobacillus rhamnosus (1x10^10 CFU/dose), Lactobacillus plantarum (4 x 10^9 CFU/dose), Bifidobacterium animalis subsp. lactis (5 x 10^9 CFU/dose), Bifidobacterium longum (1 x 10^9 CFU/dose) + 4g/dose of partially hydrolysed guar gum (PHGG).
  Mode of administration: oral.
  Interventions: Combination Product: Synbiotic
- Synbiotic + gut-directed hypnotherapy (Experimental): Includes the daily oral synbiotic (as pervious described) + a home-based therapy program.
  Home-based therapy program: based on the Manchester model of gut-directed hypnotherapy (GDH) adapted for use in children with ASD. The GDH core therapy focus areas will be relaxation, control of gut function and ego-strengthening.
  Schedule: daily use of a home-based audio recordings. The program will consist of six (6) therapy sessions/recordings over 12 weeks. Each recording (sessions 1 through 6) is to be used daily for a fortnight. Each session is approximately 15-20 minutes in duration.
  Interventions: Combination Product: Synbiotic; Behavioral: Gut-directed Hypnotherapy

INTERVENTIONS:
Combination Product: Synbiotic — Prebiotic + Probiotic
Behavioral: Gut-directed Hypnotherapy — Psychotherapy sessions
  Arms: Synbiotic + gut-directed hypnotherapy

SUMMARY:
CLINICAL ISSUE: Children with Autism Spectrum Disorder (ASD) are four times more likely to suffer with functional gastrointestinal disorders (FGIDs) than their neurotypical peers. The presence of FGIDs are linked to increased undesirable behaviour and ASD severity. Current behavioural approaches for ASD therapy do not alleviate the high comorbidity of FGIDs within this population.

BACKGROUND: Dysfunction of the microbiome-gut-brain (MGB) axis has been implicated in pathogenesis of both ASD and FGIDs. Probiotics and prebiotics can modulate the gut microbiome and research has shown efficacy at improving gastrointestinal (GI) symptoms in children with ASD and neurotypical (NT) children with FGIDs. Gut-directed hypnotherapy (GDH) has shown utility in treating FGIDs in NT children and adults but has not yet been trialed in children with ASD. Targeting therapies to address the dysfunction of the bidirectional MGB axis will likely be more effective than either brain/behavioural or gut-based therapy alone.

HYPOTHESIS: A synbiotic (prebiotic + probiotic mixture) with combined GDH will be more effective than a synbiotic alone at reducing GI symptoms in children with ASD aged 5.00 to 10.99 years over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 5.00 years to 10.99 years
2. A confirmed diagnosis of ASD or Pervasive Developmental Disorders (PDD) including autistic disorder, Asperger's disorder (AS); PDD not otherwise specified (PDD-NOS); and atypical autism.
3. A diagnosis of a functional gastrointestinal disorder (FGID) by a gastroenterologist or a score of three and above on the six-item gastrointestinal severity index (6-GSI). Accepted FGIDs include diarrhoea, constipation, bloating, abdominal pain or irritable bowel syndrome (IBS).

Exclusion Criteria:

1. Non-verbal children and/or those with severe cognitive impairment
2. Confirmed diagnosis of inflammatory bowel disease, coeliac disease, or current infection of the GI tract.

3) Any other medication, supplement or conditions which can impact the gut microbiome, including:

* antibiotics or antifungals in the last month
* probiotic or prebiotic supplements in the last two weeks
* immunocompromised or severely ill
* bipolar, schizophrenia, personality disorders
* diabetes mellitus or an eating disorder

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
GI symptom severity | Baseline, 12 weeks, 24 weeks
  Change in GI symptom severity as measured by the 6-item gastrointestinal severity index (6-GSI). The 6-GSI assesses each GI symptom using a Likert scale of 0-2 (0 = nil/mild/infrequent; 1 = moderate/occasional; 2 = severe/frequent). Score range 0-12. Mild GI issues are defined as a score of under three and moderate or severe GI issues defined as a score of three or above.

SECONDARY OUTCOMES:
ASD severity/behaviour | Baseline, 12 weeks
  Change in ASD severity scores as measured by the Aberrant Behaviour Checklist (ABC) questionnaire. The ABC consists of five subscales, including: 1) irritability (15 items); 2) lethargy/social withdrawal(16 items); 3) Stereotypic Behaviour (7 items); 4) hyperactivity/noncompliance (16 items); and 5) Inappropriate Speech (4 items). Each item is scored as 0=never a problem, 1=slight problem, 2=moderately serious problem, or 3= severe problem. The score range is 0-174, with a higher score indicating greater severity or difficulties.
Anxiety | Baseline, 12 weeks
  Change in anxiety levels as measured by the Parent Rated Anxiety Scale - Autism Spectrum Disorder (PRAS-ASD) questionnaire. This is a 25-item tool using a Likert scale of 0-3 (0=none; 1=mild; 2=moderate; 3=severe). Score range 0-75, with higher scores indicating greater levels of anxiety.
Gut microbiome | Baseline, 12 weeks
  This is an explorative outcome to compare and characterise changes in gut (stool) microbiome composition and functional profiles using shotgun metagenomic sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne K Mitchell, B.HlthSc (Hons), Principal Investigator — The University of Queensland
Locations (1):
- University of Queensland, Child Health Research Centre, Faculty of Medicine, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
IPD is the intellectual property of the funding industry partner.